CLINICAL TRIAL: NCT06857812
Title: Significance of Ultrasound Combined with Near-Infrared Spectroscopy in Monitoring Transfusion-Associated Intestinal Injury in Extremely Preterm Infants: a Study Protocol for a Prospective, Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2024531
Record Dates: First submitted 2025-02-18; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Transfusion-Associated Intestinal Injury，Ultrasound，Near-Infrared Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Extremely preterm infants: This study is an observational study with no interventions. Inclusion Criteria: 1. preterm infants with a gestational age between 23+0 and 31+6 weeks. 2. infants hospitalized in our hospital's NICU after birth, receiving a blood transfusion during hospitalization. 3. infants whose parents provide written informed consent.
  Exclusion Criteria: 1. Presence of severe congenital malformations or chromosomal abnormalities, 2. anemia due to acute blood loss; 3. presence of severe hemodynamic disorders, coagulation dysfunction, and disseminated intravascular coagulation (DIC); 4. presence of neonatal necrotizing enterocolitis, sepsis, or severe infectious conditions such as septicemia that remain uncorrected before transfusion; 5. congenital hematological diseases (such as pure red cell aplasia); 6. death due to other complications; 7. incomplete data; 8. infants participating in other interventional studies
  Interventions: Other: there is no intervention

INTERVENTIONS:
Other: there is no intervention — there is no intervention

SUMMARY:
Background: Most preterm infants with a gestational age <32 weeks in the neonatal intensive care unit (NICU) undergo blood transfusion therapy during their hospital stay to enhance their oxygen-carrying capacity and improve the oxygenation of vital organs. However, anemia and blood transfusions can lead to intestinal damage. Bedside abdominal ultrasonography and near-infrared spectroscopy (NIRS) are widely applied to monitor intestinal injury and oxygen perfusion. We hypothesized that in preterm infants (gestational age <32 weeks) with anemia and indications for transfusion, signs of intestinal injury detected by abdominal ultrasound and NIRS may appear earlier than clinical symptoms, signs, and other auxiliary examinations. Herein, we present the protocol of a study designed to assess whether abdominal ultrasonography and NIRS could therefore improve the timeliness, sensitivity, and accuracy of intestinal injury diagnosis, thereby improving prognosis.

Methods: This prospective observational study will enroll infants with a gestational age between 23+0 and 31+6 weeks with neonatal anemia, who meet the criteria for blood transfusion, and scheduled to receive transfusion therapy. In addition to routine clinical symptoms, signs, and other auxiliary examination monitoring during the transfusion process, abdominal ultrasound and NIRS findings will be analyzed. The primary outcome is the prediction intestinal injury related to anemia/transfusion using ultrasound and NIRS. A sample size of 100 cases has been set.

Conclusion: The etiology of transfusion-associated neonatal enterocolitis (TANEC) remains unclear and may result from multiple factors. Several prospective studies have assessed the significance and advantages of abdominal ultrasound combined with NIRS for monitoring intestinal injury in anemic states and transfusion therapy. Therefore, this trial aims to test the following hypothesis: monitoring intestinal injury in preterm infants (gestational age < 32 weeks) with anemia receiving red blood cell transfusions using abdominal ultrasound and NIRS can provide real-time information on changes in intestinal oxygenation during transfusion, to identify specific signs and trends in the digestive system prior to clinical symptoms and other auxiliary examination methods, thereby guiding and adjusting clinical decisions more accurately, sensitively, and rapidly. Thus, monitoring could reduce or prevent the occurrence and progression of intestinal injury, thereby improving long-term survival and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* 1. preterm infants with a gestational age between 23+0 and 31+6 weeks, 2. infants hospitalized in our hospital's NICU after birth, receiving a blood transfusion during hospitalization; and 3. infants whose parents provide written informed consent.

Exclusion Criteria:

* 1. Presence of severe congenital malformations or chromosomal abnormalities, 2. anemia due to acute blood loss; 3. presence of severe hemodynamic disorders, coagulation dysfunction, and disseminated intravascular coagulation (DIC); 4. presence of neonatal necrotizing enterocolitis, sepsis, or severe infectious conditions such as septicemia that remain uncorrected before transfusion; 5. congenital hematological diseases (such as pure red cell aplasia); 6. death due to other complications; 7. incomplete data; 8. infants participating in other interventional studies; and 8. infants whose parents do not consent to their participation.

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 100
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Abdominal Ultrasound Monitoring | abdominal ultrasound is assessed before transfusion(baseline measurement), and follow-up after transfusion Hour 0,Hour 1, Hour 2-4, Hour 6, Hour 12 , Day 1, Day 2 and Day 3.
  The infants will undergo abdominal ultrasound monitoring at fixed time points before and after transfusion. The main monitoring indicators will include the portal vein, intestinal wall structure, intestinal wall thickness, bowel width, interloop distances, bowel motility, abdominal effusion, and flow velocity/resistance index (RI) of the superior mesenteric artery (SMA).

SECONDARY OUTCOMES:
NIRS monitoring | NIRS is assessed before transfusion(baseline measurement), and follow-up after transfusion Hour 0,Hour 1, Hour 2-4, Hour 6, Hour 12 , Day 1, Day 2 and Day 3.
  Owing to the thinness and excellent penetration of the neonatal abdominal wall, the abdominal bowel oxygen saturation (regional oxygen saturation, rSO2) can be monitored using NIRS. This represents the "weighted average" of the arterial and venous partial oxygen saturation of hemoglobin in tissues approximately 1 to 2 cm deep under the sensor. The specific method is as follows: the infant is placed in a supine position, and the probe is fixed on the body surface 0.5 to 1.0 cm below the umbilicus. Except for physical examination and completion of X-ray photography, during which the probe must be removed, intestinal rSO2 will be continuously monitored using the NIRS monitor.

OTHER OUTCOMES:
clinical signs and symptoms | all assessed before transfusion(baseline measurement), and follow-up after transfusion Hour 0,Hour 1, Hour 2-4, Hour 6, Hour 12 , Day 1, Day 2 and Day 3.

IPD SHARING:
Plan to Share IPD: Yes